CLINICAL TRIAL: NCT06025851
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase I Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Escalating Intravenous Doses of CM-101 in Healthy Male Subjects
Brief Title: Intravenous Doses of CM-101 as a Treatment for Medical Conditions Involving Inflammatory and Fibrotic Mechanisms in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-I-001
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-human CCL24 monoclonal antibody (CM-101) (Experimental): Anti-human CCL24 monoclonal antibody (CM-101) Four (4) treatment groups (0.75 mg/kg, 2.5 mg/kg, 5.0 mg/kg, 10 mg/kg)
  Interventions: Drug: Anti-human CCL24 monoclonal antibody (CM-101)
- Placebo (Placebo Comparator): Placebo - intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anti-human CCL24 monoclonal antibody (CM-101) — Intravenous Infusion of Anti-human CCL24 monoclonal antibody (CM-101)
  Arms: Anti-human CCL24 monoclonal antibody (CM-101)
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
The study is designed to investigate the safety and tolerability of CM-101 for the treatment of medical conditions involving inflammatory and fibrotic mechanisms such as non-alcoholic steatohepatitis (NASH) and primary sclerosing cholangitis (PSC) and systemic sclerosis (SSc).

DETAILED DESCRIPTION:
A total of 32 male subjects were enrolled into the study and randomized to 4 treatment groups. The study was comprised of a screening period, a treatment day, a follow-up (FU) period of 42 days and an end of study (EOS) FU visit. In each Dose Group subjects was randomized to receive a single IV infusion of CM-101.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must provide written informed consent prior to participating in the study.
2. Considered healthy by the Investigator as defined by no clinically relevant abnormalities identified by a detailed medical history, full physical examination, 12-lead ECG and clinical laboratory tests.
3. Body Mass Index (BMI) 19.0-29.0 kg/m2 and total body weight within 55-95 Kg.
4. Fertile men must agree to use a barrier contraceptive (condom) for 90 days post-dosing and are restricted from donating sperm for 90 days after dosing. Subjects with a vasectomy performed more than 6 months prior to treatment are also acceptable.
5. Non-smoking and no use of any tobacco or nicotine product by declaration for a period for at least 3 month prior to screening period.
6. Supine blood pressure and heart rate within normal limits (systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 45-100 beats per minute). No evidence of orthostatic hypotension.
7. ECG with no clinically significant abnormalities recorded at Screening visit and on dosing day (before drug administration): PR interval within 120 and 210 ms, QRS interval < 120 ms, and QTc interval <450 ms.
8. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically relevant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies,). This includes any acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or CM-101 administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
2. History or current drug/alcohol abuse. History of regular alcohol consumption exceeding - 14 drinks/week for men (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening.
3. Hypereosinophilia defined as peripheral blood Eosinophils > 4.5×108/L (450/μl) or exceeding 7% of the circulating leukocytes.
4. Positive urine drug of abuse (DoA) in screening and on admission.
5. Positive breath alcohol test on admission.
6. Known acute or chronic allergy to any drug or hypersensitivity to any of the test compounds or contraindication to test product.
7. Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
8. Having received any biological treatment with recombinant antibodies, immunological therapy, or anticancer treatment. Previous standard vaccination treatment is allowed.
9. Positive HIV, hepatitis HBsAg or hepatitis HCV Ab serology tests at Screening.
10. Subjects who donated blood in the 3 months or received blood or plasma derivatives in the 6 months preceding study drug administration.
11. Participation in another clinical trial within 3 months prior to dosing (calculated from the previous study's last dosing day).
12. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of dosing, which is considered of significance by the Principal Investigator
13. Subjects with an inability to communicate well with the investigators and CRC staff (e.g., language problem, poor mental development).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Incidence and characteristics of adverse events (AEs) occurring following single doses of CM 101. | 1 day single-dose administration over 10 weeks
  Incidence and characteristics of adverse events (AEs) occurring following single doses of CM 101.
Plasma Pharmacokinetic (PK) parameters of CM-101 - Maximum CM-101 plasma concentration (Cmax) | 1 day single-dose administration over 10 weeks
  Observed maximum plasma concentration
Plasma Pharmacokinetic (PK) parameters of CM-101 - Time to Cmax (tmax) | 1 day single-dose administration over 10 weeks
  Time to reach the observed maximum plasma concentration (Tmax)
Plasma Pharmacokinetic (PK) parameters of CM-101 - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf | 1 day single-dose administration over 10 week
  Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf
Plasma Pharmacokinetic (PK) parameters of CM-101 - Terminal elimination rate constant (λz) | 1 day single-dose administration over 10 week
  Elimination rate constant, determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve
Plasma Pharmacokinetic (PK) parameters of CM-101 - Terminal elimination half-life (T½) | 1 day single-dose administration over 10 week
  Terminal elimination half-life, defined as 0.693/λz

SECONDARY OUTCOMES:
Assessment, based on the safety profile | 1 day single-dose administration over 10 week
  Assessment, based on the safety profile, whether dose-limiting toxicity (DLT) and MTD are attained within the tested doses range of CM-101.
Level of antibodies against CM-101 | 1 day single-dose administration over 10 week
  Immunogenicity as expressed by formation anti drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No